CLINICAL TRIAL: NCT04252066
Title: A Global Prospective Observational Study of Women With Fabry Disease and Their Infants During Pregnancy and Breastfeeding
Status: Recruiting | Type: Observational
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: AT1001-037
Record Dates: First submitted 2019-12-18; First posted 2020-02-05 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Fabry Disease
Keywords: migalastat; Fabry Disease; Women with Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — migalastat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1 will be pregnant and/or breastfeeding patients who have Fabry Disease, and have been exposed to at least 1 dose of migalastat during pregnancy and/or breastfeeding.
  Interventions: Drug: migalastat
- Cohort 2: Cohort 2 will be pregnant and/or breastfeeding patients who have Fabry Disease, who were not exposed to migalastat during pregnancy and/or breastfeeding.

INTERVENTIONS:
Drug: migalastat — This is an observational study. Patients as described in Cohort 1 should have been exposed to at least 1 dose of migalastat during pregnancy and/or breastfeeding.
  Groups: Cohort 1

SUMMARY:
This is a global prospective observational study of women with Fabry disease and their infants during pregnancy and/or breastfeeding. The study will evaluate outcomes of pregnancy and/or breastfeeding in women and infants exposed to migalastat.

DETAILED DESCRIPTION:
This is a global prospective observational study of women with Fabry disease and their infants during pregnancy and/or breastfeeding. The study will evaluate outcomes of pregnancy and/or breastfeeding in women and infants exposed to migalastat. All pregnant women with Fabry disease are eligible to enroll, an unexposed cohort potentially can be used for comparisons.

Cases will be reported voluntarily to the Pregnancy Coordinating Center (PCC) from any country by Healthcare Providers (HCPs), by patients and secondary contacts. The PCC will follow patients throughout their pregnancies and/or breastfeeding and infant through 1 year of age.

There will be 2 cohorts enrolled in the study. Cohort 1 will be pregnant and/or breastfeeding patients who have Fabry Disease, and have been exposed to at least 1 dose of migalastat during pregnancy and/or breastfeeding. Cohort 2 will be pregnant and/or breastfeeding patients who have Fabry Disease, who were not exposed to migalastat during pregnancy and/or breastfeeding.

This is an observational study, it will enroll patients and collect data as described in this protocol for a minimum of 10 years.

ELIGIBILITY:
Inclusion Criteria:

Female patients meeting the following criteria will be eligible for study enrollment:

1. Patients with Fabry disease who are pregnant and/or breastfeeding, whether or not they are exposed to migalastat
2. Able and willing to provide informed consent or assent, if applicable.
3. Able and willing to provide HCP contact information.

Exclusion Criteria:

None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant and/or breastfeeding patients with Fabry disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Number of major birth defects | Through the pregnancy, an average of 40 weeks and up to 12 months of infant age

SECONDARY OUTCOMES:
Incidence of spontaneous abortion | : up to 20 weeks
Number of elective or induced abortion | Through the pregnancy, an average of 40 weeks
Number of fetal death or stillbirth | Greater than 20 weeks of pregnancy and through the pregnancy, average of 40 week
Number of live birth | at the delivery, an average of 40 weeks of pregnancy
Number of neonatal death | up to 28 days of neonatal life
Number of minor birth defects | Through the pregnancy, an average of 40 weeks and up to 12 months of infant age
Number of ectopic or molar pregnancy | Through the pregnancy, an average of 40 weeks
  an ectopic or molar pregnancy occurs outside of the uterus.
Neurodevelopmental problems | Through the pregnancy, an average of 40 weeks and up to 12 months of infant age
Adverse fetal outcomes other than birth defects | Through the pregnancy, an average of 40 weeks and up to 12 months of infant age
Number of obstetric and delivery complications | At the delivery, an average of 40 weeks of pregnancy
Occurrence of Jaundice cases in Infants | Up to 1 year
Number of hospitalizations in infants | Up to 1 year
Mortality in Infants | Up to 1 year
Head circumference in Infants (cm) | Up to 1 year
Weight in Infants (kilograms) | Up to 1 year
Length in Infants (cm) | Up to 1 year
Occurrence of milk allergic reaction in breastfed or formula supplemented infants | Up to 1 year
Occurrence of allergic reaction in patients who are breastfeeding | Up to 1 year
Frequency of adverse events effecting lactation | Up to 1 year
Incidence of all serious adverse events | Through the pregnancy, an average of 40 weeks and up to 12 months of infant age

CONTACTS AND LOCATIONS:
Locations (1):
- Amicus Therapeutics, Inc. Pregnancy Registry, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No